CLINICAL TRIAL: NCT02227784
Title: The Addition of Evacetrapib to Atorvastatin Compared to Placebo, High Intensity Atorvastatin, and Atorvastatin With Ezetimibe to Evaluate LDL-C Lowering in Patients With Primary Hyperlipidemia - The ACCENTUATE Study
Brief Title: A Study of Evacetrapib (LY2484595) in Participants With High Cholesterol
Acronym: ACCENTUATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study termination due to program termination.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14502; I1V-MC-EIBH (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — evacetrapib; Atorvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atorvastatin + Evacetrapib (Experimental): Atorvastatin 40 milligrams (mg) orally once daily for 28 days during lead in period. Atorvastatin 40 mg plus evacetrapib 130 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
  Interventions: Drug: Evacetrapib; Drug: Atorvastatin; Drug: Placebo
- Atorvastatin 80 mg (Active Comparator): Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 80 mg orally with placebo for blinding once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Atorvastatin + Ezetimibe (Active Comparator): Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg plus ezetimibe 10 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe; Drug: Placebo
- Atorvastatin 40 mg (Active Comparator): Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
  Arms: Atorvastatin + Evacetrapib
Drug: Atorvastatin — Administered orally
Drug: Ezetimibe — Administered orally
  Arms: Atorvastatin + Ezetimibe
Drug: Placebo — Administered orally

SUMMARY:
The purpose of the ACCENTUATE study is to evaluate whether the study drug known as evacetrapib is effective in treating participants with high cholesterol and atherosclerotic cardiovascular disease (ASCVD) and/or diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Must be treated with atorvastatin 40 mg/day for at least 30 days prior to screening
* Have an LDL-C >70 mg/deciliter(dL) or non-HDL-C >100 mg/dL
* Have screening triglycerides ≤400 mg/dL (≤4.5 millimoles/Liter)
* Individuals with ASCVD and/or individuals with type 1 or type 2 diabetes

Exclusion Criteria:

* Have a hemoglobin A1c (HbA1c) >9.5%
* New York Heart Association (NYHA) class III or IV congestive heart failure
* History of either a transient ischemic stroke or ischemic stroke <30 days
* History of acute coronary syndrome (ACS) <30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (64):
- United States (61):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Desert Clinical Research, Mesa, Arizona
  - Central Phoenix Med Clinic LLC, Phoenix, Arizona
  - Advanced Clinical Research, Carmichael, California
  - Tooraj Joseph Raoof M.D., Inc., Encino, California
  - Irvine Clinical Research Center, Irvine, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Rancho Cucamonga Clinical, Rancho Cucamonga, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Cardiac Research, Colorado Springs, Colorado
  - ZASA Clinical Research, Boynton Beach, Florida
  - Cardiology Research Assoc., Daytona Beach, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - Alan Graff, MD, PA, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Cardiology Partners Clinical Research Institute, LLC, Wellington, Florida
  - Georgia Heart Specialists, Covington, Georgia
  - United Osteoporosis Center, Gainesville, Georgia
  - East West Medical Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - Indiana Heart Physicians Inc, Indianapolis, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Hutchinson Clinic, Hutchinson, Kansas
  - Community Medical Associates, Louisville, Kentucky
  - Grace Research, Bossier City, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Heart and Vascular Center of New Brunswick LLC, Somerset, New Jersey
  - Medex Healthcare Research, Inc., New York, New York
  - Saratoga Clinical Research LLC, Saratoga Springs, New York
  - Buffalo Cardiology and Pulmonary Associates, P.C., Williamsville, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Metrolina Internal Medicine, P.A., Charlotte, North Carolina
  - High Point Clinical Trials Center, High Point, North Carolina
  - Boice Willis Clinic, PA, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Aventiv Research, Columbus, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Portland Preventive Cardiology, LLC, Portland, Oregon
  - Partners in Clinical Research, Cumberland, Rhode Island
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Black Hills Cardiovascular Research Group, Rapid City, South Dakota
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - Northwest Houston Heart Center, Tomball, Texas
  - National Clinical Research - Richmond, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Kootenai Heart Clinics, LLC, Spokane, Washington
  - Clinical Investigation Specialists Inc, Kenosha, Wisconsin
- Puerto Rico (3):
  - Research and Cardiovascular Corp., Ponce
  - Clinical Research Puerto Rico, Inc., San Juan
  - GCM Medical Group PSC, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Nicholls SJ, Ray KK, Ballantyne CM, Beacham LA, Miller DL, Ruotolo G, Nissen SE, Riesmeyer JS; ACCENTUATE Investigators. Comparative effects of cholesteryl ester transfer protein inhibition, statin or ezetimibe on lipid factors: The ACCENTUATE trial. Atherosclerosis. 2017 Jun;261:12-18. doi: 10.1016/j.atherosclerosis.2017.04.008. Epub 2017 Apr 8. PMID 28412650

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin + Evacetrapib Open-Label (OLE): Open label extension (OLE) (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
Period: Double-Blind Phase
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe | Atorvastatin + Evacetrapib Open-Label (OLE)
Started | 123 | 54 | 62 | 127 | 0
Completed | 83 | 36 | 41 | 88 | 0
Not Completed | 40 | 18 | 21 | 39 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0
Not completed — Sponsor Decision | 34 | 15 | 14 | 32 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 5 | 2 | 0
Period: Open-Label Extension Phase (OLE)
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe | Atorvastatin + Evacetrapib Open-Label (OLE)
Started | 0 (After the double-blind treatment phase, participants entered an OLE phase.) | 0 (After the double-blind treatment phase, participants entered an OLE phase.) | 0 (After the double-blind treatment phase, participants entered an OLE phase.) | 0 (After the double-blind treatment phase, participants entered an OLE phase.) | 248 (After the double-blind treatment phase, participants entered an OLE phase.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 247
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 248
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 243
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin + Evacetrapib: Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg plus evacetrapib 130 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe | Total
Number analyzed (Participants) | 123 | 54 | 62 | 127 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.7) | 62.7 (9.3) | 61.7 (10.2) | 64.7 (8.9) | 63.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 15 | 18 | 53 | 124
  Male | 85 | 39 | 44 | 74 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 3 | 9 | 13 | 38
  Not Hispanic or Latino | 110 | 51 | 53 | 114 | 328
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 4 | 1 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 8 | 15 | 14 | 56
  White | 97 | 44 | 46 | 110 | 297
  More than one race | 3 | 1 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 123 | 54 | 62 | 127 | 366

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to 3 Months in Low-Density Lipoprotein Cholesterol (LDL-C)
Description: Change in LDL-C levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. LDL-C was measured by beta quantification. Statistics are from analysis of covariance with log baseline measurement and treatment is included in the model. Least Square Means (LS means) and median differences were analyzed in log units and converted to standard units. Log Percent change from baseline response is the dependent variable.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable LDL-C data
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | -33.44 [-34.47 to -32.41] | 0.04 [-1.01 to 1.09] | -6.19 [-7.24 to -5.15] | -27.30 [-28.33 to -26.27]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -33.48, 95% CI 2-sided [-44.4 to -23.3]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -27.24, 95% CI 2-sided [-36.6 to -18.5]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p = 0.045, ANCOVA; Median Difference (Final Values) = -6.14, 95% CI 2-sided [-12.2 to -0.22]

2. Secondary Outcome: Percent Change From Baseline to 3 Months in High-Density Lipoprotein Cholesterol (HDL-C)
Description: Change in HDL-C levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. LS medians and median differences were analyzed in log units and converted to standard units. Statistics are from mixed model repeated measures analysis with log baseline measurement, treatment, visit, and treatment by visit interaction included in the model. Log percent change from baseline response is the dependent variable. Within-participant repeated measures at multiple visits are modeled by a compound symmetry covariance structure.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable HDL-C data.
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | 125.39 [124.37 to 126.40] | 0.11 [-0.92 to 1.13] | -6.10 [-7.12 to -5.07] | -2.18 [-3.20 to -1.17]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = 125.28, 95% CI 2-sided [117.1 to 133.6]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = 131.48, 95% CI 2-sided [123.5 to 139.5]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = 127.57, 95% CI 2-sided [120.1 to 135.0]

3. Secondary Outcome: Percent Change From Baseline to 3 Months in Apolipoprotein AI (apoAI)
Description: Change in apoAI levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. Statistics are from analysis of covariance with log baseline measurement and treatment is included in the model. LS means and median differences were analyzed in log units and converted to standard units. Log Percent change from baseline response is the dependent variable.
Time Frame: Baseline, 3 Months
Population: All randomized participants with evaluable apoAI data.
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | 46.08 [45.07 to 47.09] | -0.27 [-1.29 to 0.76] | -6.14 [-7.16 to -5.12] | -2.36 [-3.38 to -1.35]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 46.35, 95% CI 2-sided [40.79 to 51.98]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 52.22, 95% CI 2-sided [47.12 to 57.33]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 48.44, 95% CI 2-sided [43.82 to 52.86]

4. Secondary Outcome: Percent Change From Baseline to 3 Months in Non-HDL-C
Description: Change in Non-HDL-C levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. LS medians and median differences were analyzed in log units and converted to standard units. Statistics are from mixed model repeated measures analysis with log baseline measurement, treatment, visit, and treatment by visit interaction included in the model. Log percent change from baseline response is the dependent variable. Within-participant repeated measures at multiple visits are modeled by a compound symmetry covariance structure.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable non-HDL-C data.
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | -31.42 [-32.44 to -30.40] | -4.95 [-5.98 to -3.92] | -9.40 [-10.44 to -8.37] | -24.37 [-25.40 to -23.35]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -26.47, 95% CI 2-sided [-33.4 to -20.0]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -22.02, 95% CI 2-sided [-28.4 to -15.9]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = -7.05, 95% CI 2-sided [-11.5 to -2.68]

5. Secondary Outcome: Percent Change From Baseline to 3 Months in Apolipoprotein B (apoB)
Description: Change in apoB levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. Statistics are from analysis of covariance with log baseline measurement and treatment is included in the model. LS means and median differences were analyzed in log units and converted to standard units. Log Percent change from baseline response is the dependent variable.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable apoB data.
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | -22.96 [-23.98 to -22.96] | 0.21 [-0.82 to 1.24] | -6.54 [-7.56 to -5.51] | -18.84 [-19.86 to -17.82]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -23.16, 95% CI 2-sided [-30.00 to -16.5]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -16.42, 95% CI 2-sided [-22.3 to -10.6]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p = 0.062, ANCOVA; Median Difference (Final Values) = -4.11, 95% CI 2-sided [-8.47 to 0.15]

6. Secondary Outcome: Percent Change From Baseline to 3 Months in Cholesterol Efflux Capacity
Description: Change in cholesterol efflux capacity from baseline to the 3-month visit expressed as a percentage of the baseline levels. Statistics are from analysis of covariance with log baseline measurement and treatment is included in the model. LS means and median differences were analyzed in log units and converted to standard units. Log Percent change from baseline response is the dependent variable.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable cholesterol efflux capacity
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin + Ezetimibe | Atorvastatin 80 mg
Number analyzed (Participants) | 86 | 40 | 44 | 91
percent | 35.09 [34.07 to 36.11] | -2.96 [-3.99 to -1.93] | -7.03 [-8.06 to -6.00] | -4.55 [-5.57 to -3.53]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 38.05, 95% CI 2-sided [30.17 to 45.88]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 42.12, 95% CI 2-sided [34.29 to 49.76]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = 39.64, 95% CI 2-sided [33.20 to 46.08]

7. Secondary Outcome: Percent Change From Baseline to 3 Months in Lipoprotein(a) (Lp[a])
Description: Change in Lp(a) levels from baseline to the 3-month visit expressed as a percentage of the baseline levels. Statistics are from analysis of covariance with log baseline measurement and treatment is included in the model. LS means and median differences were analyzed in log units and converted to standard units. Log Percent change from baseline response is the dependent variable.
Time Frame: Baseline, 3 Months
Population: All randomized participants who had evaluable Lp(a) data.
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Atorvastatin + Evacetrapib | Atorvastatin 40 mg | Atorvastatin 80 mg | Atorvastatin + Ezetimibe
Number analyzed (Participants) | 86 | 44 | 40 | 91
percent | -28.73 [-29.77 to 27.69] | 4.45 [3.40 to 5.50] | 3.90 [2.86 to 4.95] | 13.42 [12.39 to 14.45]
Statistical Analysis 1: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -33.18, 95% CI 2-sided [-44.9 to -22.3]
Statistical Analysis 2: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -32.63, 95% CI 2-sided [-44.0 to -21.8]
Statistical Analysis 3: Comparison: Atorvastatin + Evacetrapib vs Atorvastatin + Ezetimibe; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -42.15, 95% CI 2-sided [-50.9 to -33.4]

ADVERSE EVENTS:
Description: 248 randomized participants from the double-blind phase moved to open-label phase but 1 participant did not receive drug. 247 randomized participants who moved to open-label phase that received drug are part of the safety population.
Groups:
- Atorvastatin + Evacetrapib Double-Blind (DB): Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg plus evacetrapib 130 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
- Atorvastatin 40 mg DB: Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
- Atorvastatin 80 mg DB: Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 80 mg orally with placebo for blinding once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
- Atorvastatin + Ezetimibe DB: Atorvastatin 40 mg orally once daily for 28 days during lead in period. Atorvastatin 40 mg plus ezetimibe 10 mg with placebo for blinding orally once daily for 90 days. Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
- Atorvastatin + Evacetrapib Open-Label (OLE): Open label extension (atorvastatin 40 mg plus evacetrapib 130 mg) is available for compliant participants.
Arm/Group | Atorvastatin + Evacetrapib Double-Blind (DB) | Atorvastatin 40 mg DB | Atorvastatin 80 mg DB | Atorvastatin + Ezetimibe DB | Atorvastatin + Evacetrapib Open-Label (OLE)
Serious Adverse Events (participants affected / at risk) | 2/123 | 3/54 | 3/62 | 3/127 | 11/247
Other Adverse Events (participants affected / at risk) | 6/123 | 5/54 | 4/62 | 5/127 | 9/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin + Evacetrapib Double-Blind (DB) (N=123) | Atorvastatin 40 mg DB (N=54) | Atorvastatin 80 mg DB (N=62) | Atorvastatin + Ezetimibe DB (N=127) | Atorvastatin + Evacetrapib Open-Label (OLE) (N=247)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin + Evacetrapib Double-Blind (DB) (N=123) | Atorvastatin 40 mg DB (N=54) | Atorvastatin 80 mg DB (N=62) | Atorvastatin + Ezetimibe DB (N=127) | Atorvastatin + Evacetrapib Open-Label (OLE) (N=247)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1) | 3 (3) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
Early termination was due to program termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days